CLINICAL TRIAL: NCT07369271
Title: Continuous Cervical Erector Spinae Plane Block Versus Interscalene Nerve Block in Shoulder Arthroscopic Surgery- A Randomized Controlled Trial
Brief Title: Continuous Cervical Erector Spinae Plane Block Versus Interscalene Nerve Block in Shoulder Arthroscopic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-ER-114-324
Record Dates: First submitted 2026-01-08; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Arthroscopy
Keywords: Shoulder arthroscopy; postoperative pain; regional anesthesia; interscalene block; erector spinae plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous Cervical Erector Spinae Plane Block (Experimental): Participants will receive an ultrasound-guided continuous cervical erector spinae plane block with perineural catheter placement as part of a standardized multimodal analgesia regimen for shoulder arthroscopic surgery. Postoperative analgesia will be provided via continuous local anesthetic infusion through the catheter per institutional protocol.
  Interventions: Procedure: Continuous Cervical Erector Spinae Plane Block
- Continuous Interscalene Block (Active Comparator): Participants will receive an ultrasound-guided continuous interscalene block with perineural catheter placement as part of a standardized multimodal analgesia regimen for shoulder arthroscopic surgery. Postoperative analgesia will be provided via continuous local anesthetic infusion through the catheter per institutional protocol.
  Interventions: Procedure: Continuous Interscalene Block
- Single-Shot Interscalene Block (Other): Observational
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: Continuous Cervical Erector Spinae Plane Block — An ultrasound-guided cervical erector spinae plane block with catheter placement will be performed. Local anesthetic will be administered through the catheter to provide continuous postoperative analgesia according to institutional protocol as part of a standardized multimodal analgesic regimen.
  Arms: Continuous Cervical Erector Spinae Plane Block
Procedure: Continuous Interscalene Block — An ultrasound-guided interscalene block with catheter placement will be performed. Local anesthetic will be administered through the catheter to provide continuous postoperative analgesia according to institutional protocol as part of a standardized multimodal analgesic regimen.
  Arms: Continuous Interscalene Block
Procedure: No intervention — as observational group
  Arms: Single-Shot Interscalene Block

SUMMARY:
Shoulder arthroscopic surgery is associated with moderate to severe postoperative pain, which may hinder early mobilization and functional recovery. Interscalene block (ISB) is commonly used to provide effective analgesia but is frequently associated with hemidiaphragmatic paralysis due to phrenic nerve involvement. Cervical erector spinae plane block (ESPB) has been proposed as an alternative regional technique that may provide analgesia while reducing respiratory-related adverse effects. This randomized controlled trial aims to compare the analgesic efficacy and safety of cervical ESPB versus continuous ISB in patients undergoing shoulder arthroscopic surgery.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial designed to evaluate whether continuous cervical erector spinae plane block (ESPB) is non-inferior to continuous interscalene block (ISB) for postoperative pain control in adult patients undergoing elective shoulder arthroscopic surgery. Eligible participants will be allocated to one of three groups: continuous cervical ESPB, continuous ISB, or a prospective observational control group receiving standard institutional analgesia with single-shot ISB.

Randomization with allocation concealment will be applied to the two interventional groups. Patients and outcome assessors will be blinded to group allocation. All regional anesthesia techniques will be performed as part of a standardized multimodal analgesic protocol.

The primary outcome is postoperative pain intensity measured using the visual analogue scale (VAS) at 24 hours after surgery. Secondary outcomes include pain scores at additional postoperative time points, cumulative opioid consumption expressed as oral morphine equivalents, measures of functional recovery, and the incidence of block-related adverse events. Respiratory-related outcomes, including hemidiaphragmatic paralysis assessed by ultrasound, as well as motor and sensory deficits and postoperative nausea and vomiting, will also be evaluated.

Analyses of the randomized intervention groups will be conducted on an intention-to-treat basis. Data from the observational control group will be analyzed descriptively to provide reference information on usual-care outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective shoulder arthroscopic surgery

Exclusion Criteria:

* Contraindications to regional analgesia
* BMI >40
* ASA physical status IV
* history of drug or opioid abuse
* preoperative upper limb motor impairment
* postoperative ventilator support or ICU admission
* Inability to provide self-reported pain assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity within postoperative 24 hours | 2 hour, 6 hours, 12 hours, and 24 hours postoperatively
  Postoperative pain intensity will be assessed using a 0-10 visual analogue scale (VAS) at 2, 6, 12, and 24 hours after surgery.

SECONDARY OUTCOMES:
Motor blockade severity | Up to 48 hours postoperatively
  Motor blockade severity in the operated upper extremity will be assessed using a standardized muscle strength grading scale ranging from 0 to 5, where 0 indicates no muscle contraction and 5 indicates normal muscle strength.
analgesic consumption | 48 hours
  Rescue analgesic requirements and cumulative opioid consumption will be recorded and converted to oral morphine equivalent doses.
Adverse events | 7 days
  Adverse events will include postoperative nausea and vomiting, signs or symptoms of local anesthetic systemic toxicity, infection, neurologic symptoms, and catheter-related complications.
Duration of motor blockade | Up to 48 hours postoperatively
  The duration of motor blockade will be defined as the time from completion of surgery to recovery of normal motor function, defined as a muscle strength grade of 5 on the standardized 0-5 muscle strength scale, in the operated upper extremity.
Sensory blockade distribution | Up to 48 hours postoperatively
  The anatomical distribution of sensory blockade will be assessed using standardized sensory examination (e.g., response to pinprick or cold sensation) across predefined dermatomal regions of the operated upper extremity.
Duration of sensory blockade | Up to 48 hours postoperatively
  The duration of sensory blockade will be defined as the time from completion of surgery to recovery of normal sensation in the operated upper extremity, as assessed by standardized clinical sensory examination.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No